CLINICAL TRIAL: NCT05606822
Title: Endoscopic Vacuum Therapy for Anastomotic Leakage After Upper Gastrointestinal Surgery / Endoscopic Vacuum Therapy for Esophageal Perforation: A Multicenter Retrospective Cohort Study
Brief Title: Endoscopic Vacuum Therapy for Transmural Defects in the Upper Gastrointestinal Tract
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Roos Pouw, Principle Investigator, Doctor of Medicine, Doctor of Philosophy, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2021.0457
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Endoscopic Vacuum Therapy; Anastomotic Leak; Esophageal Perforation; Esophageal Perforation, Traumatic; EsoSponge; VACStent
MeSH Terms: conditions — Anastomotic Leak; Esophageal Perforation | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anastomotic leakage after gastrointestinal surgery: No interventions will be administered, as this is an observational study.
  Interventions: Other: Observational
- Esophageal perforation (Boerhaave syndrome, iatrogenic, trauma, other): No interventions will be administered, as this is an observational study.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Collection of data from electronic health record

SUMMARY:
The goal of this observational study is to learn about the best indications and techniques regarding endoscopic vacuum therapy (EVT) in patients with a transmural defect in the upper gastrointestinal (GI) tract (e.g. anastomotic leakage, Boerhaave syndrome, iatrogenic perforation, other). The main questions it aims to answer are:

* What is the success rate of EVT for transmural defects in the upper GI tract?
* What are the best indications for EVT in the upper GI tract? (e.g. etiology, patient characteristics, defect characteristics)
* What are the best techniques for EVT in the upper GI tract? (e.g. EsoSponge, VACStent, vacuum pressure, intraluminal/intracavitary) Participants will be asked for informed consent to retrospectively and prospectively collect data on EVT.

DETAILED DESCRIPTION:
Transmural defects in the upper gastrointestinal (GI) tract are defined as a disruption or injury extending through all layers of the oesophageal or gastric wall. These defects can result from various causes, including anastomotic leakage (AL) after oesophago-gastric surgery, iatrogenic perforation, Boerhaave syndrome, or trauma. Transmural defects in the upper GI tract are associated with serious consequences, such as leakage of saliva, gastric contents, and bile into the mediastinum, triggering an inflammatory response. Untreated or inadequately managed mediastinitis can lead to serious morbidity, sepsis, and mortality. Therefore, timely diagnosis and treatment of these defects is crucial. There are several treatment options for transmural defects in the upper GI tract. Conservative management involves a nil by mouth protocol, antibiotics, and (percutaneous) drainage. Endoscopic treatments include self-expandable metallic stents (SEMS), through-the-scope clips, over-the-scope clips, suturing with overstitch, and most recently, endoscopic vacuum therapy (EVT). Historically, SEMS has been the most used treatment option for transmural defects in the upper GI tract. However, persisting leakage and complications such as dislocation of the stent are not uncommon. Besides that, not all defects are suitable for stenting and additional percutaneous drainage is often necessary, but not always possible. Surgical treatment, such as a re-anastomosis or resection of the gastric conduit with construction of a cervical esophagostomy is generally required in severely septic patients. The choice of treatment depends on factors such as the location and size of the leakage, severity of symptoms, and presence of conduit ischemia or necrosis. In the past decade, EVT has been established as an effective and safe endoscopic treatment option, and it was found to be superior in terms of success rate in AL healing compared to other treatments. However, the implementation of EVT in clinical practice might be hindered by multiple challenges and questions regarding indications and techniques. This study aims to answer remaining questions and bundle expertise, to be able to determine the best indications and techniques of EVT, to reach the full potential of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treated with EVT for anastomotic leakage after esophago-gastric surgery
* Signed informed consent form
* 18 years or older

Exclusion Criteria:

* No signed informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with EVT for a transmural defect in the upper GI tract, including anastomotic leakage, Boerhaave syndrome, iatrogenic perforations, trauma, etc.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 1-3 years
  Successful treatment of EVT for the upper GI defect: closure confirmed via endoscopy

SECONDARY OUTCOMES:
Mortality | 6 months (due to possible prolonged hospital stay)
  30-day and in-hospital mortality, relation to EVT
Adverse events | 6 months
  (Severe) adverse events related to EVT
Treatment cycles | 6 months
  Including number of EVT-related endoscopies, number of used sponges/VACStents
Duration of treatment | 6 months
  Including duration of treatment in days, hospital stay in days, ICU stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Roos Pouw, MD, PhD, Principal Investigator — Amsterdam University Medical Center, location VU
Locations (1):
- Amsterdam University Medical Centers, location VUmc, Amsterdam, Netherlands

REFERENCES:
- [Derived] Pattynama LMD, Pouw RE, Henegouwen MIVB, Daams F, Gisbertz SS, Bergman JJGHM, Eshuis WJ. Endoscopic vacuum therapy for anastomotic leakage after upper gastrointestinal surgery. Endoscopy. 2023 Nov;55(11):1019-1025. doi: 10.1055/a-2102-1691. Epub 2023 May 30. PMID 37253387
- [Derived] Luttikhold J, Pattynama LMD, Seewald S, Groth S, Morell BK, Gutschow CA, Ida S, Nilsson M, Eshuis WJ, Pouw RE. Endoscopic vacuum therapy for esophageal perforation: a multicenter retrospective cohort study. Endoscopy. 2023 Sep;55(9):859-864. doi: 10.1055/a-2042-6707. Epub 2023 Feb 24. PMID 36828030
- See also: Pattynama, L. M. D. et al (2024). Multi-modality management of defects in the gastrointestinal tract: Where the endoscope meets the scalpel: Endoscopic vacuum therapy in the upper gastrointestinal tract — https://doi.org/10.1016/j.bpg.2024.101901